CLINICAL TRIAL: NCT00043329
Title: Post-Marketing Surveillance Study of Actimmune (Interferon Gamma-1b) in Patients With Severe Malignant Osteopetrosis
Brief Title: Post Marketing Surveillance Study of Actimmune in Patients With Severe, Malignant Osteopetrosis
Status: Completed | Type: Observational
Sponsor: InterMune (Industry)
Other Study IDs: GIOS-003
Record Dates: First submitted 2002-08-07; First posted 2002-08-20 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Osteopetrosis
Keywords: Registry; Actimmune; osteopetrosis
MeSH Terms: conditions — Osteopetrosis

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Drug: Actimmune Registry — as administered by physician

SUMMARY:
The purpose of this study is to establish a registry of all children with severe, malignant osteopetrosis who are treated with Actimmune (IFN-g 1b or Interferon gamma-1b) to monitor the effects of IFN-g 1b on preventing progression of this disease and to follow the safety of patients receiving it on a long-term basis. In addition, evaluation of the possible effect of Actimmune therapy on the humoral response to normal childhood vaccinations in this same patient population will be examined.Interferon gamma is a substance that the body makes naturally.

DETAILED DESCRIPTION:
It is made by white blood cells and appears to be involved in regulating the body's ability to fight off infection. Actimmune is a synthetic form of Interferon gamma which is similar to that normally made by white blood cells.

IFN-g 1b (Actimmune®) is currently approved by the United States Food and Drug Administration (FDA) for the treatment of patients with chronic granulomatous disease (CGD) to reduce the frequency and severity of serious infections. It is also approved in patients with severe, malignant osteopetrosis to delay the time to disease progression. In research trials, IFN-g 1b has been given to over 2,000 patients in diseases such as CGD, osteopetrosis, atopic dermatitis, pulmonary fibrosis, atypical mycobacteria and various cancers.

ELIGIBILITY:
* Male or female
* Diagnosis of severe, malignant osteopetrosis
* Currently receiving or planning to initiate therapy with Actimmune (Interferon gamma-1b)
* Willing to attend follow-up appointments every 6 months following enrollment into the study, if clinically indicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osteopetrosis patients receiving Actimmune therapy
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2002-01; Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Porter, MD, Study Director — InterMune
Locations (1):
- InterMune, Inc., Brisbane, California, United States